CLINICAL TRIAL: NCT00155363
Title: The Impact of Conventional Hemodialysis, High Flux Hemodialysis and Hemodiafiltration on Adiponectin, Vascular Function and Clinical Prognosis
Brief Title: Effect of Different Hemodialysis Modality on Adiponectin,Vascular Function and Clinical Prognosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9361701293
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-06

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

INTERVENTIONS:
Device: conventional artificial kidney (AK) vs. high flux AK

SUMMARY:
Adiponectin, an adipose tissue derived protein, with anti-inflammatory properties that is secreted from adipose tissue, is associated with insulin resistance. It has been shown to be a predictor of cardiovascular events in both the general population and patients undergoing hemodialysis. Adiponectin levels were inversely related to body mass index values, plasma leptin levels, insulin levels, serum triglyceride levels, and homeostatic model assessment index values. In addition to it's ability in increasing insulin sensitivity, adiponectin was demonstrated to have anti-inflammatory and anti-atherogenic properties. In patients with ESRD, renal replacement method was either peritoneal dialysis or HD. High efficient dialysis methods such as high flux HD and HDF had been used more and more popularly. High flux HD and HDF have the advantages in middle to large molecule removal, and better hemodynamic stability. Better clinical prognosis has been shown in patients undergoing high flux HD or HDF. Although studies have demonstrated that the plasma adiponectin levels were elevated in patients receiving HD, whether different dialysis modality will interfere the plasma adiponectin levels and patients' prognosis remain unknown. The current project is planned to investigate the effects of different HD modality on the plasma adiponectin levels and its correlation other serum inflammatory markers and vascular function. Patients' long term prognosis will also be assessed in the present study.

DETAILED DESCRIPTION:
Adiponectin, a cytokine with anti-inflammatory properties that is secreted from adipose tissue, is associated with insulin resistance (Horm Metab Res 34:469-474, 2002). The plasma adiponectin level has been reported to be decreased in some insulin-resistant states, such as obesity and type 2 diabetes (Biochem Biophys Res Commun 257:79-83, 1999), and coronary artery disease (CAD). However, it is shown to increase in chronic renal failure and type 1 diabetes. (European Journal of Endocrinology 148;293-300, 2003). Plasma adiponectin levels were inversely related to body mass index values, plasma leptin levels, insulin levels, serum triglyceride levels, and homeostatic model assessment index values (J Am Soc Nephrol 13:134-141, 2002, Clin Sci 103:137-142, 2002, Arterioscler Thromb Vasc Biol 20:1595-1599, 2000, Diabetes 52:942-947, 2003). In addition to it's ability in increasing insulin sensitivity, adiponectin was demonstrated to have anti-inflammatory and anti-atherogenic properties. (European Journal of Endocrinology 148;293-300, 2003, J Hypertens 18:1207-1213, 2000). It is also associated with vascular function independent of insulin sensitivity (Diabetes Care 27:739-745, 2004). In patients with ESRD, CAD remained the leading cause of death (Kidney Int 62:1417-1422, 2002) regardless of different renal replacement methods (peritoneal dialysis or HD) and the modality it uses. In recent years, with the development of high flux HD and HDF, the dialyzer has gained much progress in its efficiency. High flux HD and HDF have the advantages in middle to large molecule removal and better hemodynamic stability (Kidney Int. 66:355-66, 2004). Adiponectin, a large molecule (30kd), was not removed readily by conventional HD (Am J Kidney Dis 43:1047-1055, 2004), but it might be removed by high flux and HDF.

Due to undialyzable characteristic and decreased excretion from impaired renal function (Am J Kidney Dis 43:1047-1055, 2004, Circulation 100:2473-2476, 1999), adiponectin level is elevated in patients receiving HD and PD. Adiponectin has been shown to be a predictor of cardiovascular events in both the general population and patients undergoing HD (J Am Soc Nephrol 13:134-141, 2002) or PD (Am J Kidney Dis 43:1047-1055, 2004). Weather the elevation of adiponectin level is a protective factor of cardiovascular risk or just a reactor from inflammatory condition remains unknown. This project was aimed to study the removal efficiency of adiponectin in high flux HD and HDF and also the consequence of long term prognosis. Besides, other metabolic and inflammatory markers such as CRP, homocystine, insulin, interleukin group will be measured. Adiponectin, an adipose tissue derived protein, with anti-inflammatory properties that is secreted from adipose tissue, is associated with insulin resistance. So this project was aimed to study:

1. The removal efficiency of adiponectin in different hemodialysis modality.
2. To figure out the role of adiponectin in ESRD patients: a protective or an inflammation marker.
3. Patients' long term prognosis will be analyzed.
4. Other metabolic and inflammatory markers such as CRP, homocystine, insulin, interleukin group and their relationship with adiponectin will be investigated.
5. Vascular function will be assessed and its correlation with adiponectin levels will be studied.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis on ESRD under regular maintenance hemodialysis, no active infection, no allergy to chosen AK, informed consent acquired

Exclusion Criteria:

Not ESRD, temporary HD, active infection, during admission, allergy to chosen AK, without informed consent

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2004-09

PRIMARY OUTCOMES:
Adiponectin and inflammatory cytokines level

SECONDARY OUTCOMES:
Cardiovascular event

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Dun Wu, MD, PhD, Study Director — National Taiwan University Hospital; Pei-Lun Chu, MD, MMS, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Yun-Lin Branch, Douliu, Taiwan